CLINICAL TRIAL: NCT03306901
Title: A Randomized Multicenter Noninferiority Trial Comparing Chemoradiotherapy Versus Esophagectomy After Endoscopic Submucosal Dissection for Superficial Esophageal Squamous Cell Carcinoma (ASSURE)
Brief Title: Chemoradiotherapy Versus Esophagectomy After Endoscopic Resection for Superficial Esophageal Squamous Cell Carcinoma
Acronym: ASSURE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Hong Kwan Kim, Chief of Department of General Thoracic Surgery, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-04-074
Record Dates: First submitted 2017-09-30; First posted 2017-10-11 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Esophagectomy; Fluorouracil; Cisplatin; Radiotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors and data analysists will be blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent Chemoradiotherapy (Experimental): Patients receive 2 courses (every 3 weeks) of chemotherapy including cisplatin (45-60mg/m2) intravenously over 1 hour on day 1 and 5-fluorouracil (3,200 ~ 4,000mg/m2) intravenously for 4 to 5 days.
  Patients receive a total of 45 Gy radiation therapy (5 days a week for 5 weeks).
  Interventions: Drug: 5-fluorouracil; Drug: Cisplatin; Radiation: Radiation therapy
- Esophagectomy (Active Comparator): Patients receive surgical resection, including Ivor Lewis esophagectomy or McKeown esophagectomy and systematic lymphadenectomy.
  Interventions: Procedure: Esophagectomy

INTERVENTIONS:
Procedure: Esophagectomy — Ivor Lewis esophagectomy or McKeown esophagectomy and systematic lymphadenectomy
  Arms: Esophagectomy
Drug: 5-fluorouracil — 3,200 ~ 4,000mg/m2 intravenously for 4 to 5 days.
  Other Names: 5-FU
  Arms: Concurrent Chemoradiotherapy
Drug: Cisplatin — 45~60mg intravenously over 1 hour on day 1
  Arms: Concurrent Chemoradiotherapy
Radiation: Radiation therapy — 45 Gy irradiation (5 days a week for 5 weeks)
  Arms: Concurrent Chemoradiotherapy

SUMMARY:
This is a randomized noninferiority multicenter trial. Patients will be stratified according to the participating hospital. Patients will be randomized to one of the treatment arms.

Arm A: Patients will receive surgical resection, including Ivor Lewis esophagectomy or McKeown esophagectomy and systematic lymphadenectomy.

Arm B: Patients will receive 5-fluorouracil (5-FU) and cisplatin-based chemotherapy concurrently with radiotherapy. Patients will receive cisplatin (45~60mg/m2) intravenously over 1 hour on day 1 and receive 5-FU (3,200 ~ 4,000mg/m2) intravenously for 4 to 5 days. Treatment will repeat every 3 weeks for 2 courses. Patients will receive a total of 45 Gy irradiation (5 days a week for 5 weeks).

Patients will be followed at 3 and 6 months after randomization, then every 6 months for following 2 and half years (up to 3 years after randomization), and 4 and 5 years after randomization. After 5 years, annual follow-up is scheduled up to 10 years after randomization.

We will analyze the results primarily with the intention-to-treatment(ITT) analysis, and then secondarily with the per-protocol(PP) analysis as well.

DETAILED DESCRIPTION:
* Compare 1-year, 2-year, 3-year, 5-year, 6-year, 7-year, 8-year, 9-year, 10-year overall survival between concurrent chemoradiotherapy and esophagectomy among patients who require additional treatment for esophageal squamous cell carcinoma endoscopically resected but found to have pT1b (submucosal invasion) or lymphovascular invasion
* Compare 1-year, 2-year, 3-year, 5-year, 6-year, 7-year, 8-year, 9-year, 10-year disease-free survival between concurrent chemoradiotherapy and esophagectomy in the same study population
* Compare quality of life between concurrent chemoradiotherapy and esophagectomy in the same study population
* Compare treatment-related adverse event between concurrent chemoradiotherapy and esophagectomy in the same study population

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years and < 80 years
2. Histologically confirmed squamous cell carcinoma of the esophagus
3. Clinical stage as cT1N0M0 (AJCC/UICC 7th Edition) according to upper GI endoscopy or endoscopic ultrasound and chest computed tomography (CT) scans
4. Pathologic examination after endoscopic submucosal dissection confirmed the presence of submucosal invasion (pathologic T1b) or lymphovascular invasion
5. For participants with multiple lesions, all of them should be resected with endoscopic submucosal dissection and at least one lesion should have pathologic submucosal invasion (pT1b) or lymphovascular invasion
6. Participants has adequate hematologic function, as evidenced by an absolute neutrophil count (ANC) ≥1000/µL, hemoglobin ≥8 g/dL, and platelets ≥85,000/µL
7. Participants has adequate hepatic and renal function as defined by aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 times the upper limit of normal ; a total bilirubin ≤1.5 times the upper limit of normal ; creatinine clearance ≥ 30mL/min/1.73m2
8. Participants should agree to participate in the study and sign the informed consent form

Exclusion Criteria:

1. Cervical esophageal cancer (proximal to 20cm from incisor teeth)
2. Regional lymph node metastasis (cN+) or distant metastasis (cM1) are suspected or confirmed on chest CT scans or positron emission tomography (PET)/CT scans (Equivocal results will be regarded as no metastasis. However, it can also perform a biopsy if necessary (optional))
3. Recurrent esophageal cancer
4. Uncontrolled systemic disease which makes participants medically unfit for additional treatment (esophagectomy or concurrent chemoradiotherapy) such as congestive heart failure, interstitial lung disease, severe pulmonary emphysema or chronic renal failure
5. Gastric conduit is not available for esophageal reconstruction (ex.: previous history of gastrectomy)
6. Synchronous or metachronous multiple cancers (within the past 3 years) with the exclusion of skin cancer, well differentiated thyroid cancer, carcinoma in situ, early cancer achieving curative endoscopic resection, or low grade prostate cancer (Gleason Score≤6)

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival | 3 years from the randomization (will be assessed up to 36 months)
  defined as the time from randomization to the date of death from any cause or the last follow-up

SECONDARY OUTCOMES:
Overall survival | 1 year, 2 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years from the randomization (will be assessed up to 60 months)
  defined as the time from randomization to the date of death from any cause or the last follow-up
Disease-free survival | 1 year, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years from the randomization (will be assessed up to 60 months)
  defined as the time from randomization to the first recurrence or the date of death from any cause or the last follow-up
Quality of life (Cancer patient-specific) | Baseline, 3 months, 6 months, 1 year, 2 years, 3 years from treatment (will be assessed up to 36 months)
  assessed by EORTC QLQ C-30
Quality of life (Esophageal cancer-specific symptom) | Baseline, 3 months, 6 months, 1 year, 2 years, 3 years from treatment (will be assessed up to 36 months)
  assessed by EORTC QLQ EOS-18
Quality of life (Gastrointestinal symptom) | Baseline, 3 months, 6 months, 1 year, 2 years, 3 years from treatment (will be assessed up to 36 months)
  assessed by GSRS
Quality of life (Depression) | Baseline, 3 months, 6 months, 1 year, 2 years, 3 years from treatment (will be assessed up to 36 months)
  assessed by PHQ-9
Quality of life (Sleep disorder) | Baseline, 3 months, 6 months, 1 year, 2 years, 3 years from treatment (will be assessed up to 36 months)
  assessed by PSQI
Quality of life (Fatigue) | Baseline, 3 months, 6 months, 1 year, 2 years, 3 years from treatment (will be assessed up to 36 months)
  assessed by BFI
Treatment-related complications or adverse events | from treatment to the date of death from any cause or last follow-up (will be assessed up to 60 months)
  assessed by NCI CTCAE ver 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Hong Kwan Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (9):
- South Korea (9):
  - National Cancer Center, Goyang-si
  - Pusan National University Hospital, Pusan
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul